CLINICAL TRIAL: NCT02835482
Title: Effect of Elevated Intraocular Pressure in Glaucoma Patients During Femtolaser Cataract Surgery
Acronym: FEMTOHTO
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulties encountered with patients inclusion and femtolaser availability
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: AGC_2014-19
Record Dates: First submitted 2016-07-11; First posted 2016-07-18 (Estimated); Last update posted 2017-12-21 (Actual); Status verified 2017-12

CONDITIONS: Glaucoma; Cataract
MeSH Terms: conditions — Glaucoma; Cataract | interventions — Phacoemulsification

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Patient with glaucoma (Experimental): Patient eligible for bilateral cataract surgery, with glaucoma. Each patient is his own control. The patient is treated with femtolaser surgery for one eye and with phacoemulsification for the other eye.
  Interventions: Procedure: Femtolaser surgery; Procedure: Phacoemulsification
- Patient without glaucoma (Other): Patient eligible for bilateral cataract surgery, without glaucoma. Each patient is his own control. The patient is treated with femtolaser surgery for one eye and with the phacoemulsification for the other eye.
  Interventions: Procedure: Femtolaser surgery; Procedure: Phacoemulsification

INTERVENTIONS:
Procedure: Femtolaser surgery
Procedure: Phacoemulsification

SUMMARY:
The use of the femtosecond laser causes an increase in the intraocular pressure (IOP) between 100 mm Hg and 200 mm Hg for a period of about 80 seconds (suction phase).

If it is known that elevated IOP accelerates the degradation of retinal ganglion cells, whose axons form the optic nerve.

No data has been published to date on potential adverse effects of femtolaser cataract surgery performed in patients with glaucomatous optic neuropathy.

Since some time, spectral-domain optical coherence tomography (SD -OCT) provides a detailed analysis of ganglion cell complex (GCC) for which the loss is a marker of glaucomatous optic neuropathy. The resolution of this device, about a few microns, can detect even a tiny loss of this layer.

The investigators propose to evaluate the effects of elevated intraocular pressure in glaucoma patients undergoing femtolaser cataract surgery, studying the GCC through SD-OCT.

ELIGIBILITY:
Inclusion Criteria:

* scheduled bilateral cataract surgery
* bilateral known glaucoma confirmed at the preoperative consultation (glaucoma group) or absence of glaucoma in both eyes at confirmed the preoperative consultation (control group).

Exclusion Criteria:

* ophthalmologic pathology known other than glaucoma
* diabetes

  * untreated hypertension
  * multiple sclerosis
  * Graves' disease
  * sarcoidosis
  * patient taking toxic drug for the optic nerve and the retina
  * neurodegenerative disease
  * all general diseases that can affect the ocular structures
  * eye surgery history
  * patient's opposition to participation in the study, according to the law on research into routine care
  * absence of affiliation to social security or to universal medical coverage
  * legally protected patient
  * pregnancy or breastfeeding

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2016-04-14 (Actual); Primary Completion 2017-11-16 (Actual); Study Completion 2017-11-16 (Actual)

PRIMARY OUTCOMES:
In patient with glaucoma, measure of the thickness of the ganglion cell complex in the operated eye with femtosecond laser versus the operated eye with phacoemulsification. | within the first 3 months after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Fondation ophtalmique Adolphe de Rothschild, Paris, France